CLINICAL TRIAL: NCT01275131
Title: Randomized, Double-Blind, Pharmacokinetic (PK) and Glucodynamic (GD) Crossover Study of Continuous Subcutaneous Insulin Infusion (CSII) of Rapid Acting Insulin Analogs With and Without Recombinant Human Hyaluronidase (rHuPH20)
Brief Title: Randomized, Double-blind, Crossover, Pharmacokinetic (PK) and Glucodynamic (GD) Study of Continuous Subcutaneous Insulin Infusion (CSII) in Participants With Type 1 Diabetes Mellitus (T1DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HALO-117-105
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Results first posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Insulin analog; Type 1 diabetes mellitus; Pharmacokinetic; Glucodynamic; Phase 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Stage 1: Insulin aspart first, then insulin aspart-rHuPH20 (Active Comparator): Participants first received 0.15 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 4 days (Days 1-4; Period 1), including during a 6-hour (hr) euglycemic clamp on Days 2 and 4.
  After a 5- to 14-day washout period, participants received 0.15 U/kg insulin aspart and 5 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) (insulin aspart-rHuPH20) coadministered as a CSII, for 4 days (Days 5-8; Period 2), including during a 6-hr euglycemic clamp on Days 6 and 8.
  Interventions: Drug: Insulin aspart; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
- Stage 1: Insulin aspart-rHuPH20 first, then insulin aspart (Active Comparator): Participants first received 0.15 units per kilogram (U/kg) insulin aspart and 5 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) (insulin aspart-rHuPH20) coadministered as a continuous subcutaneous insulin infusion (CSII), for 4 days (Days 1-4; Period 1), including during a 6-hour (hr) euglycemic clamp on Days 2 and 4.
  After a 5- to 14-day washout period, participants received 0.15 U/kg insulin aspart alone as a CSII, for 4 days (Days 5-8; Period 2), including during a 6-hr euglycemic clamp on Days 6 and 8.
  Interventions: Drug: Insulin aspart; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
- Stage 3: Insulin aspart first, then insulin aspart + rHuPH20 (Active Comparator): Participants first received 0.12 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 5 days (Days 1-5; Period 1), including during a 6-hour (hr) euglycemic clamp on Days 2, 3, and 5. On Day 2 only, a sham injection was administered 2.5 hr prior to the 6-hr euglycemic clamp.
  After a 5- to 14-day washout period, participants received 0.12 U/kg insulin aspart administered as a CSII, for 5 days (Days 6-10; Period 2), including during a 6-hr euglycemic clamp on Days 7, 8, and 10. On Day 7 only, a 1.0-milliliter (mL) subcutaneous (SC) injection of 1.25 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) was administered 2.5 hr prior to the 6-hr euglycemic clamp.
  Interventions: Drug: Insulin aspart; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
- Stage 3: Insulin aspart + rHuPH20 first, then insulin aspart (Active Comparator): Participants first received 0.12 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 5 days (Days 1-5; Period 1), including during a 6- hour (hr) euglycemic clamp on Days 2, 3, and 5. On Day 2 only, a 1.0-milliliter (mL) subcutaneous (SC) injection of 1.25 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) was administered 2.5 hr prior to the euglycemic clamp .
  After a 5- to 14- day washout period, participants received 0.12 U/kg insulin aspart administered as a CSII, for 5 days (Days 6-10; Period 2), including during a 6-hr euglycemic clamp on Days 7, 8, and 10. On Day 7 only, a sham injection was administered 2.5 hr prior to the 6-hour euglycemic clamp.
  Interventions: Drug: Insulin aspart; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)

INTERVENTIONS:
Drug: Insulin aspart
  Other Names: Novolog
Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
  Other Names: PH20; Hylenex

SUMMARY:
The purpose of this study is to determine if recombinant human hyaluronidase PH20 (rHuPH20) will change the exposure and action of approved insulin analogs when given by continuous subcutaneous insulin infusion (CSII) in participants with Type 1 diabetes mellitus (T1DM).

This study is divided into Stage 1, 2, and 3. Stage 3 was started chronologically before Stage 2 and, prior to performing Stage 2, the Sponsor made the decision to terminate Stage 2. Stage 2 was not initiated due to a strategic business decision and termination was not based on safety or efficacy concerns. No participants were enrolled in Stage 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 65 years, inclusive. Females of child-bearing potential must use a standard and effective means of birth control for the duration of the study.
2. Non-smoking participants with Type 1 diabetes mellitus (T1DM) treated with insulin for greater than or equal to 12 months. Non-smoking means abstinence from cigarettes and cigars for 3 months and negative cotinine screening tests.
3. Body mass index (BMI) 18.0 to 35.0 kilograms per meter squared (kg/m^2), inclusive.
4. Glycosylated hemoglobin A1c (HbA1c) ≤10 % based on local laboratory results.
5. Fasting C-peptide <0.6 nanograms per milliliter (ng/mL).
6. Current treatment with insulin <90 units per day (U/d).
7. Routine use of continuous subcutaneous insulin infusion (CSII) as the primary route of insulin administration.
8. Participant should be in good general health based on medical history and physical examination, without medical conditions that might prevent the completion of study drug infusions and assessments required in this protocol.

Exclusion Criteria:

1. Known or suspected allergy to any component of any of the study drugs in this trial.
2. Previous enrollment in this trial (Exception: participants in Stage 1 are permitted to participate in Stage 2).
3. Use of drugs that may interfere with the interpretation of trial results or are known to cause clinically relevant interference with insulin action, glucose utilization, or recovery from hypoglycemia. Participants taking maintenance doses of blood thinners (eg, Coumadin or heparin) will be excluded.
4. Use of any long-acting insulin injection within 72 hours of Stage 1 or Stage 3.
5. Recurrent major hypoglycemia or hypoglycemic unawareness, as judged by the Investigator.
6. Current addiction to alcohol or substances of abuse as determined by the Investigator.
7. Blood donation or phlebotomy (>500 milliliters [mL]) within the previous 8 weeks of Screening. This applies both to new participants and to participants who have participated in Stage 1 and who wish to continue in Stage 2.
8. Pregnancy, breast-feeding, the intention of becoming pregnant, or not using adequate contraceptive measures (adequate contraceptive measures consist of sterilization, intra-uterine device [IUD], oral or injectable contraceptives, or barrier methods).
9. Symptomatic gastroparesis.
10. Receipt of any investigational drug within 4 weeks of Stage 1 or Stage 2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Morrow, MD, Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (1):
- Profil Institute for Clinical Research, Chula Vista, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1: Insulin Aspart First, Then Insulin Aspart-rHuPH20: Participants first received 0.15 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 4 days (Days 1-4; Period 1), including during a 6-hour (hr) euglycemic clamp on Days 2 and 4.
  After a 5- to 14-day washout period, participants received 0.15 U/kg insulin aspart and 5-micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) (insulin aspart-rHuPH20) coadministered as a CSII, for 4 days (Days 5-8; Period 2), including during a 6-hr euglycemic clamp on Days 6 and 8.
- Stage 3: Insulin Aspart First, Then Insulin Aspart + rHuPH20: Participants first received 0.12 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 5 days (Days 1-5; Period 1), including during a 6-hour (hr) euglycemic clamp on Days 2, 3, and 5. On Day 2 only, a sham injection was administered 2.5 hr prior to the 6-hr euglycemic clamp.
  After a 5- to 14-day washout period, participants received 0.12 U/kg insulin aspart administered as a CSII, for 5 days (Days 6-10; Period 2), including during a 6-hr euglycemic clamp on Days 7, 8, and 10. On Day 7 only, a 1.0 milliliter (mL) subcutaneous (SC) injection of 1.25 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) was administered 2.5 hr prior to the 6-hr euglycemic clamp.
- Stage 3: Insulin Aspart + rHuPH20 First, Then Insulin Aspart: Participants first received 0.12 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 5 days (Days 1-5; Period 1), including during a 6-hour (hr) euglycemic clamp on Days 2, 3, and 5. On Day 2 only, a 1.0 milliliter (mL) subcutaneous (SC) injection of 1.25 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) was administered 2.5 hr prior to the 6-hr euglycemic clamp .
  After a 5- to 14-day washout period, participants received 0.12 U/kg insulin aspart administered as a CSII, for 5 days (Days 6-10; Period 2), including during a 6-hr euglycemic clamp on Days 7, 8, and 10. On Day 7 only, a sham injection was administered 2.5 hr prior to the 6-hr euglycemic clamp.
Period: Period 1
Arm/Group | Stage 1: Insulin Aspart First, Then Insulin Aspart-rHuPH20 | Stage 1: Insulin Aspart-rHuPH20 First, Then Insulin Aspart | Stage 3: Insulin Aspart First, Then Insulin Aspart + rHuPH20 | Stage 3: Insulin Aspart + rHuPH20 First, Then Insulin Aspart
Started | 11 | 9 | 13 | 12
Received at Least One Dose of Study Drug | 11 | 9 | 13 | 12
Completed | 9 | 9 | 10 | 10
Not Completed | 2 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 0
Period: 5- to 14-Day Washout Period
Arm/Group | Stage 1: Insulin Aspart First, Then Insulin Aspart-rHuPH20 | Stage 1: Insulin Aspart-rHuPH20 First, Then Insulin Aspart | Stage 3: Insulin Aspart First, Then Insulin Aspart + rHuPH20 | Stage 3: Insulin Aspart + rHuPH20 First, Then Insulin Aspart
Started | 9 | 9 | 10 | 10
Completed | 9 | 9 | 10 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Period 2 (Crossover)
Arm/Group | Stage 1: Insulin Aspart First, Then Insulin Aspart-rHuPH20 | Stage 1: Insulin Aspart-rHuPH20 First, Then Insulin Aspart | Stage 3: Insulin Aspart First, Then Insulin Aspart + rHuPH20 | Stage 3: Insulin Aspart + rHuPH20 First, Then Insulin Aspart
Started | 9 | 9 | 10 | 10
Completed | 8 | 8 | 9 | 8
Not Completed | 1 | 1 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Stage 1: Insulin Aspart First, Then Insulin Aspart-rHuPH20: Participants first received 0.15 units per kilogram (U/kg) insulin aspart, administered as a continuous subcutaneous insulin infusion (CSII), for 4 days (Days 1-4; Period 1), including during a 6-hour (hr) euglycemic clamp on Days 2 and 4.
  After a 5- to 14-day washout period, participants received 0.15 U/kg insulin aspart and 5 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) (insulin aspart-rHuPH20) coadministered as a CSII, for 4 days (Days 5-8; Period 2), including during a 6-hr euglycemic clamp on Days 6 and 8.
- Stage 3: Insulin Aspart First, Then Insulin Aspart + rHuPH20: Participants first received 0.12 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 5 days (Days 1-5; Period 1), including during a 6-hour (hr) euglycemic clamp on Days 2, 3, and 5. On Day 2 only, a sham injection was administered 2.5 hr prior to the 6-hr euglycemic clamp.
  After a 5- to 14-day washout period, participants received 0.12 U/kg insulin aspart administered as a CSII for 5 days (Days 6-10; Period 2), including during a 6-hr euglycemic clamp on Days 7, 8, and 10. On Day 7 only, a 1.0-milliliter (mL) subcutaneous (SC) injection of 1.25 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) was administered 2.5 hr prior to a 6-hr euglycemic clamp.
- Stage 3: Insulin Aspart + rHuPH20 First, Then Insulin Aspart: Participants first received 0.12 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 5 days (Days 1-5; Period 1), including during a 6-hour (hr) euglycemic clamp on Days 2, 3, and 5. On Day 2 only, a 1.0-milliliter (mL) subcutaneous (SC) injection of 1.25 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) was administered 2.5 hr prior to the euglycemic clamp .
  After a 5- to 14-day washout period, participants received 0.12 U/kg insulin aspart administered as a CSII, for 5 days (Days 6-10; Period 2), including during a 6-hr euglycemic clamp on Days 7, 8, and 10. On Day 7 only, a sham injection was administered 2.5 hr prior to a 6-hr euglycemic clamp.
- Total: Total of all reporting groups
Arm/Group | Stage 1: Insulin Aspart First, Then Insulin Aspart-rHuPH20 | Stage 1: Insulin Aspart-rHuPH20 First, Then Insulin Aspart | Stage 3: Insulin Aspart First, Then Insulin Aspart + rHuPH20 | Stage 3: Insulin Aspart + rHuPH20 First, Then Insulin Aspart | Total
Number analyzed (Participants) | 11 | 9 | 13 | 12 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.3 (6.39) | 44.6 (9.00) | 35.5 (9.50) | 32.3 (10.29) | 35.44 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 7 | 6 | 22
  Male | 5 | 6 | 6 | 6 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 2
  White | 11 | 9 | 11 | 11 | 42
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 10 | 8 | 13 | 12 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 11 | 9 | 13 | 12 | 45

OUTCOME MEASURES:

1. Primary Outcome: Early Insulin Exposure (%AUC[0-60]), Stage 1
Description: Early insulin exposure, defined as the percentage of total insulin exposure (area under the insulin concentration curve [AUC{0-360}]) that occurs within the first hour following bolus dose of insulin during the 2 euglycemic clamps is presented. Blood samples were collected 10 minutes predose and at 0, 5, 10, 15, 20, 30, 45, 60, 120, 150, 180, 240, 300, and 360 minutes postdose during the euglycemic clamp.
Time Frame: 10 minutes predose up to 60 minutes postdose
Population: Participants who completed all study periods within a given stage with evaluable early insulin exposure (%AUC[0-60]) data.
Measure: Mean (Standard Deviation); unit: Percentage of AUC(0-360)
Groups:
- Stage 1: Insulin Aspart Alone: Participants received 0.15 units per kilogram (U/kg) insulin aspart, administered as a continuous subcutaneous insulin infusion (CSII), for 4 days (Days 1-4 or 5-8), including during a 6-hour (hr) euglycemic clamp on Days 2 and 4 of Period 1 or Days 6 and 8 of Period 2
- Stage 1: Insulin Aspart-rHuPH20: Participants received 0.15 units per kilogram (U/kg) insulin aspart and 5 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) (insulin aspart-rHuPH20) coadministered as a continuous subcutaneous insulin infusion (CSII), for 4 days (Days 1-4 or 5-8), including during a 6-hour (hr) euglycemic clamp on Days 2 and 4 of Period 1 or Days 6 and 8 of Period 2
Arm/Group | Stage 1: Insulin Aspart Alone | Stage 1: Insulin Aspart-rHuPH20
Number analyzed (Participants) | 16 | 16
Percentage of AUC(0-360)
  Stage 1, Day 2/6 | 20.99 (6.37) | 34.94 (9.48)
  Stage 1, Day 4/8 | 32.83 (14.66) | 50.97 (13.91)
Statistical Analysis 1: Comparison: Stage 1: Insulin Aspart Alone vs Stage 1: Insulin Aspart-rHuPH20; Comparison at Stage 1, Day 2/6; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; A mixed model with fixed effects for treatment, day, and interaction of treatment with day was performed using a compound symmetric covariance matrix; Least Squares Mean Difference = 13.95, 90% CI 2-sided [7.37 to 20.54]
Statistical Analysis 2: Comparison: Stage 1: Insulin Aspart Alone vs Stage 1: Insulin Aspart-rHuPH20; Comparison at Stage 1, Day 4/8; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = 18.14, 90% CI 2-sided [11.55 to 24.72]

2. Secondary Outcome: Maximum Glucose Infusion Rate (GIRmax), Stage 1
Description: Maximum glucose infusion rates (GIRmax) for Stage1 are presented. Blood samples were collected at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 0 up to 360 minutes postdose on Day 2/6 and Day 4/8
Population: Participants who completed all periods of study within a given stage with evaluable GIRmax data.
Measure: Mean (Standard Deviation); unit: Milligrams/kilogram/minute
Groups:
- Stage 1: Insulin Aspart Alone: Participants received 0.15 units per kilogram (U/kg) insulin aspart, administered as a continuous subcutaneous insulin infusion (CSII), for 4 days (Days 1-4 or 5-8), including during a 6-hour (hr) euglycemic clamp on Days 2 and 4 of Period 1 or Day 6 and 8 of Period 2.
- Stage 1: Insulin Aspart-rHuPH20: Participants received 0.15 units per kilogram (U/kg) insulin aspart and 5 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) (insulin aspart-rHuPH20) administered together as a continuous subcutaneous insulin infusion (CSII), for 4 days (Days 1-4 or 5-8), including during a 6-hour (hr) euglycemic clamp on Days 2 and 4 of Period 1 or Days 6 and 8 of Period 2.
Arm/Group | Stage 1: Insulin Aspart Alone | Stage 1: Insulin Aspart-rHuPH20
Number analyzed (Participants) | 16 | 16
Milligrams/kilogram/minute
  Stage 1, Day 2/6 | 13.37 (4.23) | 12.51 (3.19)
  Stage 1, Day 4/8 | 11.88 (3.64) | 11.52 (3.67)

3. Primary Outcome: Early Exposure to Insulin (%AUC[0-60]), Stage 3
Description: Early insulin exposure, defined as the percentage of total insulin exposure (area under the insulin concentration curve [AUC{0-360}) that occurs within the first hour following bolus dose of insulin during the 2 euglycemic clamps is presented. Blood samples were collected 10 minutes predose and at 0, 5, 10, 15, 20, 30, 45, 60, 120, 150, 180, 240, 300, and 360 minutes postdose during the euglycemic clamp.
Time Frame: 10 minutes predose up to 60 minutes postdose on Days 2/7, 3/8, and 5/10
Population: Participants who completed all periods of study within a given stage with evaluable %AUC(0-60) data.
Measure: Mean (Standard Deviation); unit: Percentage of AUC(0-360)
Groups:
- Stage 3: Insulin Aspart Alone: Participants received 0.12 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 5 days (Days 1-5 or 6-10), including during a 6-hour (hr) euglycemic clamp on Days 2, 3, and 5 of Period 1, or on Days 7, 8, and 10 of Period 2. On Day 2 or Day 7 only, a sham injection was administered 2.5 hr prior to the 6-hr euglycemic clamp.
- Stage 3: Insulin Aspart + rHuPH20: Participants received 0.12 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 5 days (Days 1-5 or 6-10), including during a 6-hour (hr) euglycemic clamp on Days 2, 3, and 5 of Period 1, or on Days 7, 8, and 10 of Period 2. On Day 2 or Day 7 only, a 1 milliliter (mL) subcutaneous (SC) injection of 1.25 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) was administered 2.5 hr prior to the 6-hr euglycemic clamp.
Arm/Group | Stage 3: Insulin Aspart Alone | Stage 3: Insulin Aspart + rHuPH20
Number analyzed (Participants) | 17 | 17
Percentage of AUC(0-360)
  Stage 3, Day 2/7 | 15.70 (6.38) | 32.11 (10.91)
  Stage 3, Day 3/8 | 22.29 (5.43) | 36.39 (9.43)
  Stage 3, Day 5/10 | 27.31 (10.49) | 32.64 (11.32)
Statistical Analysis 1: Comparison: Stage 3: Insulin Aspart Alone vs Stage 3: Insulin Aspart + rHuPH20; Comparison at Stage 3, Day 2/7; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed model with fixed effects for treatment, day, and interaction of treatment with day. A compound symmetric covariance matrix was assumed; Least Squares Mean Difference = 16.41, 90% CI 2-sided [11.86 to 20.97]
Statistical Analysis 2: Comparison: Stage 3: Insulin Aspart Alone vs Stage 3: Insulin Aspart + rHuPH20; Comparison at Stage 3, Day 3/8; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Least Squares Mean Difference = 14.10, 90% CI 2-sided [9.55 to 18.65]
Statistical Analysis 3: Comparison: Stage 3: Insulin Aspart Alone vs Stage 3: Insulin Aspart + rHuPH20; Comparison at Stage 3, Day 5/10; Test type: Superiority or Other; p = 0.0552, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Least Squares Mean Difference = 5.32, 90% CI 2-sided [0.77 to 9.88]

4. Secondary Outcome: Maximum Glucose Infusion Rate (GIRmax), Stage 3
Description: Maximum glucose infusion rates (GIRmax) for Stage 3 are presented. Blood samples were collected at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 0 up to 360 minutes postdose on Days 2/7, 3/8, and 5/10
Population: Participants who completed all periods of study within a given stage with evaluable GIRmax data.
Measure: Mean (Standard Deviation); unit: Milligrams/kilogram/minute
Groups:
- Stage 3: Insulin Aspart Alone: Participants received 0.12 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 5 days (Days 1-5 or 6-10), including during a 6-hour (hr) euglycemic clamp on Days 2, 3, and 5 of Period 1, or Days 7, 8, and 10 of Period 2. On Day 2 or Day 7 only, a sham injection was administered 2.5 hr prior to the 6-hr euglycemic clamp.
- Stage 3: Insulin Aspart + rHuPH20: Participants received 0.12 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 5 days (Days 1-5 or 6-10), including during a 6-hour (hr) euglycemic clamp on Days 2, 3, and 5 of Period 1, or on Days 7, 8, and 10 of Period 2. On Day 2 or Day 7 only, a 1-milliliter (mL) subcutaneous (SC) injection of 1.25 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) was administered 2.5 hr prior to the 6-hr euglycemic clamp.
Arm/Group | Stage 3: Insulin Aspart Alone | Stage 3: Insulin Aspart + rHuPH20
Number analyzed (Participants) | 17 | 17
Milligrams/kilogram/minute
  Stage 3, Day 2/7 | 9.58 (2.28) | 12.63 (3.88)
  Stage 3, Day 3/8 | 10.07 (3.36) | 12.4 (3.39)
  Stage 3, Day 5/10 | 9.97 (3.53) | 10.76 (3.35)

5. Secondary Outcome: Time to First Occurrence of Maximum Glucose Infusion Rate (tGIRmax), Stage 1
Description: Time to first occurrence of maximum glucose infusion rate (tGIRmax) for Stage 1 is presented. Blood samples were collected at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 0 up to 360 minutes postdose on Day 2/6 and Day 4/8
Population: Participants who completed all periods of study within a given stage with evaluable tGIRmax data.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Stage 1: Insulin Aspart Alone | Stage 1: Insulin Aspart-rHuPH20
Number analyzed (Participants) | 16 | 16
Minutes
  Stage 1, Day 2/6 | 115.38 (59.21) | 102.38 (38.28)
  Stage 1, Day 4/8 | 92.50 (24.71) | 84.31 (25.89)

6. Secondary Outcome: Time to First Occurrence of Maximum Glucose Infusion Rate (tGIRmax), Stage 3
Description: Time to first occurrence of maximum glucose infusion rate (tGIRmax) for Stage 3 is presented. Blood samples were collected at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 0 up to 360 minutes postdose on Days 2/7, 3/8, and 5/10
Population: Participants who completed all periods of study within a given stage with evaluable tGIRmax data.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Stage 3: Insulin Aspart Alone | Stage 3: Insulin Aspart + rHuPH20
Number analyzed (Participants) | 17 | 17
Minutes
  Stage 3, Day 2/7 | 127.65 (60.02) | 78.53 (27.04)
  Stage 3, Day 3/8 | 135.24 (73.00) | 79.47 (42.57)
  Stage 3, Day 5/10 | 117.76 (75.20) | 79.53 (42.99)

7. Secondary Outcome: Time to 50% Maximum Glucose Infusion Rate (tGIR50%Max), Stage 1
Description: Early and late times to 50% maximum glucose infusion rate (tGIR50%max) for Stage 1 are presented. Blood samples were collected at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 0 up to 360 minutes postdose on day 2/6 and Day 4/8
Population: Participants who completed all periods of study within a given stage with evaluable early or late tGIR50%max data.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Stage 1: Insulin Aspart-rHuPH20: Participants received 0.15 units per kilogram (U/kg) insulin aspart and 5 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) (insulin aspart-rHuPH20) administered together as a continuous subcutaneous insulin infusion (CSII), for 4 days, including during a 6-hour (hr) euglycemic clamp on Days 2 and 4 or Days 6 and 8.
Arm/Group | Stage 1: Insulin Aspart Alone | Stage 1: Insulin Aspart-rHuPH20
Number analyzed (Participants) | 16 | 16
Minutes
  Early tGIR50%max, Stage 1, Day 2/6 | 46.50 (18.08) | 34.88 (17.92)
  Late tGIR50%max, Stage 1, Day 2/6 | 162.19 (56.78) | 158.06 (52.58)
  Early tGIR50%max, Stage 1, Day 4/8 | 35.19 (28.54) | 39.75 (18.71)
  Late tGIR50%max, Stage 1, Day 4/8 | 132.63 (47.37) | 114.19 (29.05)

8. Secondary Outcome: Time to 50% Maximum Glucose Infusion Rate (tGIR50%Max), Stage 3
Description: Early and late time to 50% maximum glucose infusion rates (tGIR50%max) for Stage 3 studies are presented. Blood samples were collected at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 0 up to 360 minutes postdose on Days 2/7, 3/8, and 5/10
Population: Participants who completed all periods of study within a given stage with evaluable early and late tGIR50%max data.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Stage 3: Insulin Aspart Alone: Participants received 0.12 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 5 days (Days 1-5 or 6-10), including during a 6 hour (hr) euglycemic clamp on Days 2, 3, and 5 of Period 1, or Days 7, 8, and 10 of Period 2. On Day 2 or Day 7 only, a sham injection was administered 2.5 hr prior to the 6-hr euglycemic clamp.
Arm/Group | Stage 3: Insulin Aspart Alone | Stage 3: Insulin Aspart + rHuPH20
Number analyzed (Participants) | 17 | 17
Minutes
  Early tGIR50%max, Stage 3, Day 2/7 | 58.47 (17.53) | 31.06 (20.73)
  Late tGIR50%max, Stage 3, Day 2/7 | 144.18 (61.44) | 98.71 (39.87)
  Early tGIR50%max, Stage 3, Day 3/8 | 32.59 (22.88) | 31.53 (21.27)
  Late tGIR50%max, Stage 3, Day 3/8 | 153.41 (65.35) | 102.88 (44.57)
  Early tGIR50%max, Stage 3, Day 5/10 | 27.29 (18.40) | 28.88 (21.97)
  Late tGIR50%max, Stage 3, Day 5/10 | 136.88 (73.39) | 110.59 (55.10)

9. Secondary Outcome: Time to 50% Total Glucose Infused (50%Gtot), Stage 1
Description: Time to 50% total glucose infused (50%Gtot) is presented for Stage 1. Blood samples were collected at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 0 up to 360 minutes postdose on Day 2/6 and Day 4/8
Population: Participants who completed all periods of study within a given stage with evaluable 50%Gtot data.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Stage 1: Insulin Aspart Alone | Stage 1: Insulin Aspart-rHuPH20
Number analyzed (Participants) | 16 | 16
Minutes
  Stage 1, Day 2/6 | 156.13 (18.70) | 134.94 (18.28)
  Stage 1, Day 4/8 | 137.38 (22.21) | 115.25 (14.50)

10. Secondary Outcome: Time to 50% Total Glucose Infused (50%Gtot), Stage 3
Description: Time to 50% of total glucose infused (50%Gtot) is presented for Stage 3. Blood samples were collected at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 0 up to 360 minutes postdose on Days 2/7, 3/8, and 5/10
Population: Participants who completed all periods of study within a given stage with evaluable 50%Gtot data.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Stage 3: Insulin Aspart Alone | Stage 3: Insulin Aspart + rHuPH20
Number analyzed (Participants) | 17 | 17
Minutes
  Stage 3, Day 2/7 | 174.59 (25.86) | 124.18 (22.03)
  Stage 3, Day 3/8 | 154.06 (24.02) | 120.00 (17.12)
  Stage 3, Day 5/10 | 146.59 (28.63) | 130.18 (23.54)

11. Secondary Outcome: Area Under the Glucose Concentration Curve (AUC[0-360]), Stage 1
Description: Area under the glucose concentration curve for 0 to 360 minutes (AUC[0-360]) from Stage 1 is presented. Blood samples were collected 30 and 10 minutes prior to insulin bolus and at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 30 minutes predose up to 360 minutes postdose on Day 2/6 and Day 4/8
Population: Participants who completed all periods of study within a given stage with evaluable AUC(0-360) data.
Measure: Mean (Standard Deviation); unit: Picomoles*minutes/liter
Arm/Group | Stage 1: Insulin Aspart Alone | Stage 1: Insulin Aspart-rHuPH20
Number analyzed (Participants) | 16 | 16
Picomoles*minutes/liter
  Stage 1, Day 2/6 | 1978.08 (631.89) | 1977.02 (795.79)
  Stage 1, Day 4/8 | 1598.40 (546.00) | 1324.31 (500.04)

12. Secondary Outcome: Area Under the Glucose Concentration Curve (AUC[0-360]), Stage 3
Description: Area under the glucose concentration curve from 0 to 360 minutes (AUC[0-360]) for Stage 3 studies is presented. Blood samples were collected 30 and 10 minutes prior to insulin bolus and at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 30 minutes predose up to 360 minutes postdose Days 2/7, 3/8, and 5/10
Population: Participants who completed all periods of study within a given stage with evaluable AUC(0-360) data.
Measure: Mean (Standard Deviation); unit: Picomoles*minutes/liter
Arm/Group | Stage 3: Insulin Aspart Alone | Stage 3: Insulin Aspart + rHuPH20
Number analyzed (Participants) | 17 | 17
Picomoles*minutes/liter
  Stage 3, Day 2/7 | 1197.60 (385.44) | 1509.38 (541.45)
  Stage 3, Day 3/8 | 1368.81 (424.16) | 1405.75 (516.85)
  Stage 3, Day 5/10 | 1289.22 (486.03) | 1369.97 (462.78)

13. Secondary Outcome: Duration of Insulin Action (AUMC[0-360]/AUC[0-360]), Stage 1
Description: Duration of insulin action was calculated by dividing the area under the first moment curve (AUMC[0-360]) by the area under the concentration versus time curve (AUC[0-360]) for Stage 1. Blood samples were collected 10 minutes predose and at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 10 minutes predose up to 360 minutes postdose on Day 2/6 and Day 4/8
Population: Participants who completed all periods of study within a given stage with evaluable AUMC(0-360)/AUC(0-360) data.
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Stage 1: Insulin Aspart Alone: Participants received 0.15 units per kilogram (U/kg) insulin aspart, administered as a continuous subcutaneous insulin infusion (CSII), for 4 days (Days 1-4 or 5-8), including during a 6 hour (hr) euglycemic clamp on Days 2 and 4 of Period 1 or Days 6 and 8 of Period 2.
Arm/Group | Stage 1: Insulin Aspart Alone | Stage 1: Insulin Aspart-rHuPH20
Number analyzed (Participants) | 16 | 16
Ratio
  Stage 1, Day 2/6 | 163.63 (14.70) | 146.51 (16.30)
  Stage 1, Day 4/8 | 147.50 (23.86) | 132.60 (15.55)

14. Secondary Outcome: Duration of Insulin Action (AUMC[0-360]/AUC[0-360]), Stage 3
Description: Duration of insulin action was calculated by dividing the area under the first moment curve (AUMC[0-360]) by the area under the concentration versus time curve (AUC[0-360]) for Stage 3. Blood samples were collected 10 minutes predose and at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 10 minutes predose up to 360 minutes postdose on Days 2/7, 3/8, and 5/10
Population: Participants who completed all periods of study within a given stage with evaluable AUMC(0-360)/AUC(0-360) data.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Stage 3: Insulin Aspart Alone | Stage 3: Insulin Aspart + rHuPH20
Number analyzed (Participants) | 17 | 17
ratio
  Stage 3, Day 2/7 | 180.39 (18.72) | 138.59 (18.41)
  Stage 3, Day 3/8 | 164.65 (19.97) | 135.71 (17.30)
  Stage 3, Day 5/10 | 156.14 (26.38) | 145.81 (16.42)

ADVERSE EVENTS:
Description: AEs were classified by the body system affected.
Groups:
- Stage 1: Insulin Aspart: Participants received 0.15 units per kilogram (U/kg) insulin aspart, administered as a continuous subcutaneous insulin infusion (CSII), for 4 days (Days 1-4 or 5-8), including during a 6-hour (hr) euglycemic clamp on Days 2 and 4 of Period 1 or Days 6 and 8 of Period 2.
- Stage 3: Insulin Aspart: Participants received 0.12 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 5 days (Days 1-5 or 6-10), including during a 6-hour (hr) euglycemic clamp on Days 2, 3 and 5 of Period 1 or Days 7, 8, and 10 of Period 2. On Day 2 or Day 7 only, a sham injection was administered 2.5 hr prior to the 6-hr euglycemic clamp.
- Stage 3: Insulin Aspart + rHuPH20: Participants received 0.12 units per kilogram (U/kg) insulin aspart administered as a continuous subcutaneous insulin infusion (CSII), for 5 days (Days 1-5 or 6-10), including during a 6-hour (hr) euglycemic clamp on Days 2, 3, and 5 of Period 1 or Days 7, 8, and 10 of Period 2. On Day 2 or Day 7 only, a 1-milliliter (mL) subcutaneous (SC) injection of 1.25 micrograms per milliliter (μg/mL) recombinant human hyaluronidase PH20 (rHuPH20) was administered 2.5 hr prior to the 6-hr euglycemic clamp.
Arm/Group | Stage 1: Insulin Aspart | Stage 1: Insulin Aspart-rHuPH20 | Stage 3: Insulin Aspart | Stage 3: Insulin Aspart + rHuPH20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 16/20 | 13/18 | 14/23 | 12/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: Insulin Aspart (N=20) | Stage 1: Insulin Aspart-rHuPH20 (N=18) | Stage 3: Insulin Aspart (N=23) | Stage 3: Insulin Aspart + rHuPH20 (N=22)
Injection site erythema (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Infusion site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infusion site oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (7) | 3 (3) | 4 (5) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vessel puncture site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion site haematoma (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Infusion site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other